CLINICAL TRIAL: NCT02857166
Title: Phase IA Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Recombinant Humanized Anti-PD-1 Monoclonal Antibody (JS001) in Patients With Advanced Solid Tumors
Brief Title: Study of JS001 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-ZSZL-I
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Solid Tumors
Keywords: JS001; solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- humanized anti-PD-1 monoclonal antibody toripalimab (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 0.3mg/kg or 1mg/kg or 3mg/kg or 10mg/kg until disease progresses or unacceptable tolerability occurs.
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody toripalimab

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody toripalimab — humanized anti-PD-1 monoclonal antibody (JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance and Dose-Limiting Toxicity (DLT) of Recombinant humanized anti-PD-1 monoclonal antibody (JS001) in patients with advanced solid tumors.

DETAILED DESCRIPTION:
OVERVIEW

This is a Phase 1, open-label, dose-escalation study of JS-001, a humanized monoclonal IgG4 antibody targeting the Programmed Death -1 (PD-1). It is estimated that 12-24 subjects with advanced or recurrent solid tumors or will be enrolled in the study.

A 3+3 design will be utilized for this Phase 1 study. Four dose levels are planned and include: 0.3, 1, 3, 10 mg/kg/dose. Each of the 4 dose levels will use 2 dose schedules: single dose, repeated doses every 2 weeks. Subjects will be assigned to a dose schedule in the order of study entry.

The study will be the traditional 3 + 3 design with 3 or 6 subjects treated at this dose level and at all subsequent dose levels depending upon the incidence of DLTs. If no DLTs occur in a cohort of 3 subjects, a new cohort of 3 subjects will be treated at the next higher dose level. If 1 of 3 subjects in a cohort experiences a DLT, that cohort will be expanded to 6 subjects. If only 1 of the 6 subjects has a DLT, then the next cohort of 3 subjects will be treated at the next higher dose level. If 2 or more DLTs occur within a cohort, then that dose level will be above the MTD (the highest dose where no more than 1 of 6 subjects has experienced a DLT), and the previous lower (tolerated) dose level will be considered the MTD.

A DLT is defined as a Grade 3 drug-related adverse event occurring within the first cycle (28 days) of dosing (excluding tumor flare defined as local pain, irritation, or rash localized at sites of known or suspected tumor or a transient Grade 3 infusion adverse event) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 in a single dose cohort.

Tumor response will be evaluated using immune-related response criteria (irRC), WHO criteria , Response Evaluation Criteria in Solid Tumors (RECIST), immune-related RECIST, and International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphomas (for lymphomas only).

In the absence of confirmed disease progression and intolerable toxicities, subjects in the single dose cohorts and multiple dose cohorts will be allowed to continue JS-001 administration with the consent of the subject.

DOSAGE AND ADMINISTRATION

JS-001 will be administered as a 60-minute i.v. infusion. Cohorts will include escalating dose levels of 0.3, 1, 3, 10mg/kg/dose.

SAFETY EVALUATIONS

Assessment of safety will be determined by vital sign measurements, clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status evaluations, diagnostic imaging, physical examinations, electrocardiograms, and the incidence and severity of adverse events.

Safety will also include evaluations of immune safety and immunogenicity. Particular attention will be given to adverse events that may follow enhanced T-cell activation such as dermatitis and colitis, uveitis, or other immune-related adverse events (irAEs).

An irAE is a clinically significant adverse event of any organ that is associated with drug exposure, of unknown etiology, and is consistent with an immune-mediated mechanism.

EFFICACY EVALUATIONS

The primary efficacy endpoint is the best response rate (RR). Duration of response, progression-free survival, time to progression, and overall survival will also be analyzed.

PHARMACOKINETIC EVALUATIONS

Pharmacokinetic parameters include AUC, Cmax, tmax, and t½, etc. STATISTICAL METHODS The sample size for this study is not determined from power analysis. It is based on the 3+3 design for dose escalation and safety evaluation requirements.

Descriptive statistics will include: mean, standard deviation, median, and minimum and maximum values for continuous variables; frequencies and percentages for categorical variables.

The efficacy parameters will be summarized using descriptive statistics. All safety and pharmacokinetic parameters will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of advanced or recurrent adenocarcinoma of solid tumor, including adenocarcinoma of the stomach or gastro-esophageal junction, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, cholangiocarcinoma, Pancreatic ductal cell carcinoma, etc.

   * at least one prior chemotherapy regimen
   * age between 18 and 75 years, both gender
   * has at least one measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST V1.1)
2. life expectancy ≥ 3 months
3. ECOG performance status of 0 or 1
4. Has had last dose of chemotherapy more than 4 weeks prior to the first dose of study therapy JS001, and has recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 Grade 1 or better from the AEs due to the chemotherapy.
5. Has had last administration of radioactive therapy more than 4 weeks prior to the first dose of study therapy JS001.
6. Has had last administration of immunosuppressive systemic steroid therapy (more than 10 mg/d prednisone or equal dose) more than 2 weeks prior to the first dose of study therapy JS001.
7. Has undergone major surgery that needs general anesthesia more than 4 weeks prior to the first dose of study therapy JS001. Has undergone surgery that needs local anesthesia or epidural anesthesia more than 72 hours prior to the first dose of study therapy JS001 and has already recovered from the surgery. Has undergone biopsy more than 1 hour prior to the first dose of study therapy JS001.
8. The lab examination results of the screening must fulfill all of the following:

   * absolute neutrophil count more than or equal to 1.5×109/ L
   * platelet count more than or equal to 90×109/ L
   * hemoglobin more than or equal to 90 g/L
   * creatinine less than or equal to132.6µmol/L or creatinine clearance >40 mL/min
   * aspartate transferase(AST) and alanine transferase(ALT) less than or equal to 3.0 ×ULN
   * total bilirubin less than or equal to 1.5×ULN( except for the patients with Gilbert syndrome, whose total bilirubin ,must less than or equal to 51.3µmol/L)
9. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to participation in any study related activities.
10. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Has had antineoplastic herbal therapy within 2 weeks prior to the first dose of study therapy JS001.
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and receive study therapy or used an investigational device within 4 weeks of the first dose of study drug.
3. Has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication.
4. Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the participant has undergone potentially curative therapy with no evidence of that disease for 5 years.
5. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. Has interstitial lung disease OR has had a history of pneumonitis that has required oral or IV steroids.
7. Has active or suspected autoimmune disease except leukoderma,type I Diabetes, Residual hypothyroidism that induced by autoimmune thyroiditis and only requires the use of hormone replacement therapy, Or disease that rarely relapse without external stimulating factors.
8. Had prior treatment targeting PD-1: anti-PD-1,anti-PD-L1, anti-PD-L2, cytotoxic T-lymphocyte-associated protein (CTLA), or other antibodies that targeting T cell costimulatory pathway or checkpoint.
9. Has an active infection requiring systematic therapy.
10. Is positive for Human Immunodeficiency Virus (HIV).
11. Has active Tuberculosis.
12. Has known active Hepatitis B or C.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
14. Has received or will receive a live vaccine within 30 days prior to the first administration of study drug.
15. Is pregnant or breastfeeding.
16. Cannot tolerate vein puncture and / or venous access.
17. Any other conclusive medical reasons, mental illness, and / or social reasons that determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Up to 2 approximately years

SECONDARY OUTCOMES:
Anti-Drug Antibody of JS001 in Chinese patients | Cycle 1,2,3,5 Day 1 before JS001 infusion and 336 hours after last JS001 infusion, each cycle is 28 days.
Objective Response Rate (ORR) | Up to 2 approximately years
Duration of Response (DOR) | Up to 2 approximately years
Progression-Free survival (PFS) | Up to 2 approximately years
Overall Survival (OS) | Up to 2 approximately years
DLT in patients with solid tumor treated with JS001. | Cycle 1（each cycle is 28 days）
PD-1 receptor occupancy of blood | 1 year
Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) | 1 year
Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb | 1 year
Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb Area Under the Curve [AUC]). Area Under the Curve (AUC) after single dose injection of Recombinant Humanized Anti-PD-1 Monoclonal Antibody | 1 year
t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb | 1 year
Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb | 1 year
Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb | 1 year
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb | 1 year
Average Plasma Concentration (Cav) of steady state after multiple dose injection of Anti-PD-1 mAb | 1 year
Degree of fluctuation (DF) of steady state after multiple dose injection of Anti-PD-1 mAb | 1 year
Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen UniversityCancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No